CLINICAL TRIAL: NCT05205863
Title: A Phase 1/2 Study of the Dose-Response in Pharmacodynamics and Safety of Prothrombin Complex Concentrate Cofact in Healthy Subjects Under Vitamin K Antagonist Anticoagulation.
Brief Title: Dose-Response in PD and Safety of Cofact Under VKA Anticoagulation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD2021.01
Record Dates: First submitted 2021-12-23; First posted 2022-01-25 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — prothrombin complex concentrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cofact Dose 1 (Experimental)
  Interventions: Biological: Cofact
- Cofact Dose 2 (Experimental)
  Interventions: Biological: Cofact
- Placebo (Placebo Comparator)
  Interventions: Biological: Cofact

INTERVENTIONS:
Biological: Cofact — Human prothrombin complex concentrate

SUMMARY:
This is a randomized, open label, placebo-controlled, parallel design, single center, prospective study. Subjects will receive treatment with VKA. Subjects who reach the targeted INR, will receive single dose of Cofact. Multiple coagulation laboratory tests will be evaluated over a period of 15 days

ELIGIBILITY:
Inclusion Criteria:

* Male or female of nonchildbearing potential.
* Healthy subjects.

Exclusion Criteria:

* Evidence of coagulation disturbances, or disposition for thrombo-embolic events
* Liver function tests more than 1.2 times the upper normal limits
* Participants with thyroid disorders as evidenced by assessment of TSH levels outside the normal reference range at screening.
* Prior history of thromboembolic complications including those in first degree relatives.
* Glomerular filtration rate (GFR) is lower than estimated GFR 62 mL/min/1.73 m2 using the Modification of Diet in Renal Disease Study equation.
* Anaphylactic or systemic reactions to human plasma, plasma products, or blood products.
* History of hypersensitivity to active or inactive excipients of VKA
* Gastrointestinal disease that may impair VKA absorption..
* Participation in another clinical study <30 days prior to study entry.
* Any clinically significant history of or current clinically significant disease or disorder as judged by the Investigator.
* Positive nasopharyngeal PCR test for SARS-CoV-2 on Day -11 or Day -1.
* Positive pregnancy test at screening, Day -11, or Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-09-03 (Actual)

PRIMARY OUTCOMES:
Peak thrombin generation at 30 minutes after end of the Cofact infusion | 30 minutes post Cofact infusion

SECONDARY OUTCOMES:
Changes in ETP | 24 hours post Cofact infusion
  Change in endogenous thrombin potential (ETP) over 24 hours after the EOI
Concentration in clotting factors | up to Day 15
  Changes in aPTT, PT, and INR
Coagulation markers | up to Day 15
  Concentration over time of clotting factors: FII, FVII, FIX, FX, protein C, and protein S
Coagulation activation markers | up to Day 15
  Concentration over time of Prothrombin fragment 1+2, D-dimer, and thrombin-antithrombin complexes (TATs)
Safety outcome | up to Day 15
  Frequency and severity of adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Salah Hadi, MD, Principal Investigator — PRA Health Sciences; Thomas Bodewes, MD, Study Chair — Prothya Biosolutions
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No